CLINICAL TRIAL: NCT01970995
Title: A Randomized, Controlled, Multi-center Study to Demonstrate Reductions in Exposure to Selected Smoke Constituents in Smokers Switching to THS 2.2 Menthol or Smoking Abstinence Compared to Smoking Menthol Conventional Cigarettes, for 90 Days
Brief Title: Reduced Exposure Study Using THS 2.2 Menthol With 5 Days in a Confinement Setting and 85 Days in an Ambulatory Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZRHM-REXA-07-JP; ZRHM-REXA-07-JP (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2013-10-18; First posted 2013-10-28 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: Candidate modified risk tobacco product; Conventional cigarettes; Reduced exposure; HPHCs; Ambulatory
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- THS 2.2 Menthol (mTHS 2.2) (Experimental): Ad libitum use of THS 2.2 Menthol for 5 Days in a Confinement Setting and 85 Days in an Ambulatory Setting
  Interventions: Other: THS 2.2 Menthol (mTHS 2.2)
- Smoking abstinence (SA) (Active Comparator): Abstinence from smoking for 5 Days in a Confinement Setting and 85 Days in an Ambulatory Setting
  Interventions: Other: Smoking Abstinence (SA)
- Menthol Conventional Cigarette (mCC) (Active Comparator): Ad libitum use of subject's own preferred brand of mCC for 5 Days in a Confinement Setting and 85 Days in an Ambulatory Setting
  Interventions: Other: Menthol Conventional Cigarette (mCC)

INTERVENTIONS:
Other: THS 2.2 Menthol (mTHS 2.2) — THS 2.2 Menthol ad libitum for 5 days in confinement prolonged by 85 days in an ambulatory setting
  Arms: THS 2.2 Menthol (mTHS 2.2)
Other: Smoking Abstinence (SA) — SA for 5 days in confinement prolonged by 85 days in an ambulatory setting
  Arms: Smoking abstinence (SA)
Other: Menthol Conventional Cigarette (mCC) — Subject's own preferred brand of mCC ad libitum for 5 days in confinement prolonged by 85 days in an ambulatory setting
  Arms: Menthol Conventional Cigarette (mCC)

SUMMARY:
The main goal of the study is to evaluate if the ad libitum use of the THS 2.2 Menthol (mTHS 2.2) for 5 days in confinement and after 85 days of product use in an ambulatory setting, by Japanese adult healthy smokers results in a reduction in the levels of biomarkers of exposure for selected harmful and potentially harmful smoke constituents (HPHCs) compared to smokers continuing smoking their own preferred brand of menthol conventional cigarette (mCC) and smoking abstinence (SA). Smokers who remained abstinent from SA were used as a benchmark to provide context to the exposure reduction.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Japanese.
* Smoking, healthy subject as judged by the Investigator.
* Subject smokes at least 10 commercially available mCCs per day (no brand restrictions) for the last 4 weeks, based on self-reporting.
* Subject has smoked for at least the last 3 consecutive years.
* Subject does not plan to quit smoking in the next 3 months.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* The subject has received medication within 14 days or within 5 half-lives of the medication (whichever is longer) which has an impact on cytochrome P450 1 A2 (CYP1A2) or cytochrome P450 2 A6 (CYP2A6) activity.
* For women: Subject is pregnant or is breast feeding.
* For women: Subject does not agree to use an acceptable method of effective contraception.

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Endo, MD, Principal Investigator — Osaki Hospital Tokyo Heart Center; Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (1):
- Osaki Hospital Tokyo Heart Center, 5-4-12, Kitashinagawa, Shinagawa-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject screened): 01 August 2013
  At admission (Day -2), all the subjects performed a product trial of the THS 2.2 Menthol. During the baseline period, they continued smoking their single preferred brand of mCC. Then, on Day 0, they were randomized to one of the 3 study arms (mTHS 2.2, mCC or SA) in a 2:1:1 ratio.
Pre-assignment Details: Enrolled and randomized population = 160 subjects
  * 78 subjects in mTHS 2.2
  * 42 subjects in mCC
  * 40 subjects in SA
  Number of subjects enrolled but NOT randomized (who tried the mTHS 2.2 at Day -2) = 0
Period: Confinement Period (Population at Day 5)
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Started | 78 | 42 | 40
Completed | 77 | 41 | 39
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Period: End of Study (Population at Day 90)
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Started | 77 | 41 | 39
Completed | 76 | 41 | 38
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study population = all randomized subjects who had at least one post randomization product use experience and at least one valid biomarker of exposure measurement.
  160 randomized subjects: 78 in mTHS 2.2, 42 in mCC and 40 in SA arms
  155 completed, subjects who withdrew: 2 in mTHS 2.2, 1 in mCC and 2 in SA arms
Groups:
- Total: Total of all reporting groups
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA) | Total
Number analyzed (Participants) | 78 | 42 | 40 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.58) | 37.4 (11.23) | 37.0 (9.96) | 37.2 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 17 | 18 | 68
  Male | 45 | 25 | 22 | 92
Daily mCC consumption at Screening [Number; unit: participants]
  10 to 19 cig/day | 40 | 23 | 21 | 84
  > 19 cig/day | 38 | 19 | 19 | 76

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Monohydroxybutenyl Mercapturic Acid (MHBMA)
Description: Concentrations measured at Day 5 in urine, adjusted for creatinine.
  Geometric Least Squares (LS) means are provided as descriptive statistics.
Time Frame: 5 days
Population: The analysis was performed on the Per Protocol set (PP) which included all randomized subjects who had no major protocol deviation impacting the evaluability during the confinement period.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 76 | 42 | 39
pg/mg creat | 83.21 [73.51 to 94.19] | 617.04 [521.87 to 729.55] | 83.57 [70.32 to 99.32]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); The hypothesis to be tested is that the geometric mean level on Day 5 of the biomarker of exposure for mTHS 2.2 is lower relative to mCC. Analysis of the biomarker of exposure (BoExp) was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 5 for mTHS 2.2 and mCC respectively; Test type: Superiority or Other; p < .001, ANCOVA — The primary endpoints were tested using a multiple testing procedure to preserve the overall alpha level by simultaneously testing the endpoints using a closed procedure with each test performed at an alpha level of 2.5% one sided; ANCOVA model on MHBMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 13.49, 95% CI 2-sided [10.96 to 16.60] — Geometric LS mean ratio mTHS 2.2:mCC

2. Primary Outcome: Concentration of 3-hydroxypropylmercapturic Acid (3-HPMA)
Description: as for outcome 1
Time Frame: 5 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mg creat
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 76 | 42 | 39
ng/mg creat | 304.56 [283.22 to 327.50] | 601.11 [545.07 to 662.91] | 183.61 [165.93 to 203.18]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); The hypothesis to be tested is that the geometric mean level on Day 5 of the biomarker of exposure for mTHS 2.2 is lower relative to mCC. Analysis of the BoExp was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 5 for mTHS 2.2 and mCC respectively; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on 3-HPMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 50.67, 95% CI 2-sided [44.88 to 57.20] — Geometric LS mean ratio mTHS 2.2:mCC

3. Primary Outcome: Concentration of S-phenylmercapturic Acid (S-PMA)
Description: as for outcome 1
Time Frame: 5 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 76 | 42 | 39
pg/mg creat | 119.18 [107.73 to 131.85] | 1086.89 [948.47 to 1245.51] | 104.83 [91.07 to 120.66]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on S-PMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 10.97, 95% CI 2-sided [9.26 to 12.99] — Geometric LS mean ratio mTHS 2.2:mCC

4. Primary Outcome: Levels of Carboxyhemoglobin (COHb)
Description: % COHb blood measurements performed in the evening of Day 5, expressed as % of saturation of hemoglobin.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 5 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: % of saturation of hemoglobin
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 76 | 42 | 39
% of saturation of hemoglobin | 2.47 [2.37 to 2.57] | 5.49 [5.21 to 5.79] | 2.49 [2.35 to 2.63]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on COHb levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 44.94, 95% CI 2-sided [42.11 to 47.97] — Geometric LS mean ratio mTHS 2.2:mCC

5. Primary Outcome: Concentration of Total 4-(Methylnitrosamino)-1-(3- Pyridyl)-1-butanol) (Total NNAL)
Description: Concentrations measured at Day 90 in urine, adjusted for creatinine.
  Geometric Least Squares (LS) means are provided as descriptive statistics.
Time Frame: 90 days
Population: The analysis was performed on the Per Protocol set (PP) which included all randomized subjects who had no major protocol deviation impacting the evaluability during the period Day 60 to Day 90.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 70 | 41 | 37
pg/mg creat | 22.48 [18.82 to 26.84] | 96.65 [76.63 to 121.90] | 14.90 [11.67 to 19.02]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); The hypothesis to be tested is that the geometric mean level on Day 90 of the biomarker of exposure for mTHS 2.2 is lower relative to mCC. Analysis of the BoExp was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 90 for mTHS 2.2 and mCC respectively; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on Total NNAL levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 23.25, 95% CI 2-sided [17.38 to 31.11] — Geometric LS mean ratio mTHS 2.2:mCC

ADVERSE EVENTS:
Time Frame: From the informed consent form signature until the end of the safety follow-up period, up to 150 days (including a screening period of up to 28 days, a 9-day confinement period followed by a 85-day ambulatory setting, and by a 28-day safety follow-up period (28 days after discharge of the subject or early discontinuation)).
Description: The safety was assessed in the safety population, consisting of 160 subjects: 160 randomized subjects (78 in mTHS 2.2, 42 in mCC and 40 in SA) and no subject exposed to mTHS 2.2 from the product trial on Day -2 but not randomized.
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 16/78 | 4/42 | 4/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THS 2.2 Menthol (mTHS 2.2) (N=78) | Menthol Conventional Cigarette (mCC) (N=42) | Smoking Abstinence (SA) (N=40)
Haemoglobin decreased (Investigations) | 11 (13) | 3 (5) | 3 (4)
Neutrophil count decreased (Investigations) | 5 (5) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specifies that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belongs to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2014-04-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT01970995/Prot_000.pdf
  • Statistical Analysis Plan (2014-11-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT01970995/SAP_001.pdf